CLINICAL TRIAL: NCT05286151
Title: Subcortical Network Connectivity and Temporal Processing in Children With Persistent and Recovered Stuttering
Brief Title: Network Connectivity and Temporal Processing in Adolescents Who Stutter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Soo-Eun Chang, Associate Professor of Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00196133; 2R01DC011277 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Stuttering, Childhood; Stuttering
Keywords: Rhythm; Temporal processing; Healthy children; Speech disorders; Timing
MeSH Terms: conditions — Stuttering; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children who stutter (Experimental): Children who stutter
  Interventions: Behavioral: Rhythm discrimination
- Children who do not stutter (Experimental): Children who do not stutter
  Interventions: Behavioral: Rhythm discrimination

INTERVENTIONS:
Behavioral: Rhythm discrimination — Participants will complete a rhythm discrimination task once per year for 3 years.

SUMMARY:
The specific purpose of this clinical trial is to compare performance on rhythm perception and production tasks between children who stutter and children who do not stutter. The overall project also aims to investigate how performance on rhythm tasks may be related to brain activity (non-clinical trial).

DETAILED DESCRIPTION:
Participants in the clinical trial portion of this study will complete rhythm discrimination and finger tapping experiments once a year for 3 years. The study team will compare performance between groups. Participants will also participate in the non-trial portion of the project that includes having magnetic resonance imaging (MRI) each year for 3 years.

ELIGIBILITY:
Inclusion Criteria Children who stutter:

* English as primary language
* Current or past stuttering diagnosis

Inclusion Criteria Children who do not stutter:

* English as primary language

Exclusion Criteria Children who stutter:

* Diagnosed/under treatment for any neurological or psychiatric conditions
* Head trauma with loss of consciousness
* Major medical illness
* Hearing loss- Language/motor delay (below -2 standard deviations on standardized assessments)
* Face, motor, or reflex abnormalities

Exclusion Criteria Children who do not stutter:

* Personal or family history of stuttering
* Diagnosed/under treatment for any neurological or psychiatric conditions
* Head trauma with loss of consciousness
* Major medical illness
* Hearing loss
* Language/motor delay (below -2 standard deviations on standardized assessments
* Face, motor, or reflex abnormalities

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2022-07-23 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Rhythm discrimination (d') | Year 1
  Performance on the rhythm discrimination task will be assessed using a signal detection analysis to distinguish between participants' ability to discriminate same and different rhythms from any general tendency to respond same or different. Hit rates (HRs) and false alarm rates (FARs) will be obtained to calculate d' (a measure of sensitivity; determined by z(HR) - z(FAR)).
Rhythm discrimination (d') | Year 2
  Performance on the rhythm discrimination task will be assessed using a signal detection analysis to distinguish between participants' ability to discriminate same and different rhythms from any general tendency to respond same or different. Hit rates (HRs) and false alarm rates (FARs) will be obtained to calculate d' (a measure of sensitivity; determined by z(HR) - z(FAR)).
Rhythm discrimination (d') | Year 3
  Performance on the rhythm discrimination task will be assessed using a signal detection analysis to distinguish between participants' ability to discriminate same and different rhythms from any general tendency to respond same or different. Hit rates (HRs) and false alarm rates (FARs) will be obtained to calculate d' (a measure of sensitivity; determined by z(HR) - z(FAR)).

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Eun Chang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No